CLINICAL TRIAL: NCT06917534
Title: The Cognitive Neural Mechanisms and Neuroregulatory Interventions of Realistic Creative Problem-solving Under the Effects of Drug Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yifan Wang (Other)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Sponsor-Investigator, Yifan Wang, Laboratory Manager, Shaanxi Normal University
Organization: Shaanxi Normal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: L20230122; 32471114 (Other Grant/Funding Number: The National Natural Science Foundation of China grant)
Record Dates: First submitted 2025-03-24; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Drug Addiction
Keywords: heroin; creative problem solving; divergent thinking; group problem solving
MeSH Terms: conditions — Substance-Related Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): The study was sham-controlled, randomized, and double-blind. Participants with HUD were randomly assigned to either the active or sham groups. The DC-STIMULATOR PLUS (neuroConn, Germany) was used to deliver stimulation via saline-soaked sponge electrodes (25 cm², 5×5 cm, 1.5 mA). The stimulation in the active group lasted for 20 min with a 30-s fade-in and a 30-s fade-out. They received five stimulation sessions within one week, with a minimum interval of 24 hours between each session. The tDCS sensitivity questionnaire was used to assess blinding validity.
  Interventions: Device: Transcranial direct current stimulation
- Sham group (Sham Comparator): Arm Description: The study was sham-controlled, randomized, and double-blind. Participants with HUD were randomly assigned to either the active or sham groups. The DC-STIMULATOR PLUS (neuroConn, Germany) was used to deliver stimulation via saline-soaked sponge electrodes (25 cm², 5×5 cm, 1.5 mA). The stimulation in the sham group was set up as a stimulation cycle of 30s fade-in and 30s fade-out, followed by no current stimulation. They received five stimulation sessions within one week, with a minimum interval of 24 hours between each session. The tDCS sensitivity questionnaire was used to assess blinding validity.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — The participant cohort recruited for this study consists of individuals with drug addiction specifically those addicted to drugs. During the intervention phase, this group will adhere to a strict non-pharmacological intervention protocol, meaning they will not receive any form of pharmacotherapy, neurosurgical intervention, or other neuromodulation-based cognitive interventions, including but not limited to techniques such as transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS). This design aims to ensure the internal validity of the study results and to exclude potential confounding effects of other interventions on neuroplasticity and cognitive function.

SUMMARY:
Drug addiction persists as a significant global social concern with a negative impact on social harmony and stability that cannot be ignored. After returning to society, individuals with drug addiction often suffer from impaired creative problem-solving abilities and difficulties in interpersonal cooperation. The difficulties in survival stress and the sense of helplessness triggered by these factors are important reasons that lead them to seek drugs repeatedly and even to commit criminal behaviors. Therefore, enhancing creative realistic problem-solving abilities emerges as a pivotal pathway for drug addicts to facilitate rehabilitation from drug addiction and achieve societal adaptation. The project emphasizes both individual and collaborative creative solution generation for realistic problem solving. The abnormal cognitive neural mechanisms and interpersonal neural mechanisms will be systematically explored by using multiple cognitive and neuroimaging methods, such as functional near-infrared spectroscopy (fNIRS), electroencephalography (EEG), and eye-tracking. From the cognitive-behavioral-brain level, a comprehensive neurophysiological multimodal predictive model of how drug addiction affects creative realistic problem-solving will be constructed by multi-level data fitting modeling. Building upon this research foundation, The investigators will further implement single and repeated sessions of transcranial direct current stimulation (tDCS) targeting damaged brain regions for the intervention of individual and collaborative problem-solving ability under the effect of drug addiction. The indicators of brain, cognition, and behavior will be tracked at multiple time points.

ELIGIBILITY:
Inclusion Criteria:

* age between 30 and 60 years;
* fulfilling the diagnostic criteria for severe substance use disorder as specified in the Fifth Edition of the Diagnostic and Statistical Manual of Mental Disorders.
* a history of heroin use exceeding ten years, with a daily average intake of at least 0.1 grams.
* abstinence duration of eight months or less, with a positive result of a urine test before entering the rehabilitation center.
* no history of neuromodulation treatments such as tDCS within the past six months.

Exclusion Criteria:

* a history of alcohol dependence, neurological disorders, or other complex psychiatric conditions.
* the presence of intracranial metallic implants or elevated intracranial pressure.
* a history of epilepsy or recent electroencephalogram evidence of epileptiform activity.
* the use of implanted electronic devices, such as pacemakers;.
* scalp hyperalgesia or a tendency toward bleeding.
* severe cardiac conditions.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Score on the Realistic Presented Problem Task | From enrollment to the end of treatment at 1 month
  Used to measure problem-solving ability individual creative problem-solving
Score on the Group Realistic Problem Solving Task | From enrollment to the end of treatment at 1 month
  Used to measure collaborative problem-solving ability
Cortical activation from fNIRS | From enrollment to the end of treatment at 1 month
Cortical functional connectivity from fNIRS | From enrollment to the end of treatment at 1 month
Inter-brain neural synchronization from fNIRS hyperscaning | From enrollment to the end of treatment at 1 month
Pupil response from eye-tracking | From enrollment to the end of treatment at 1 month
Score on the Alternative Use Task | From enrollment to the end of treatment at 1 month
  Used to measure the individual problem-solving ability
Score on the Group Alternative Use Task | From enrollment to the end of treatment at 1 month
  Used to measure collaborative problem-solving

SECONDARY OUTCOMES:
Average fixation duration from eye-traking | From enrollment to the end of treatment at 1 month
Fixation time percentage from eye-traking | From enrollment to the end of treatment at 1 month
Score on the joint drawing task | From enrollment to the end of treatment at 1 month
  Used to measure collaborative problem-solving from the perspective of social interaction.
Score on the Chain Free Association Task | From enrollment to the end of treatment at 1 month
  Used to measure remote associative ability.
Score on the Verbal Fluency Task | From enrollment to the end of treatment at 1 month
  Used to measure remote association ability
Score on the Divergent Association Task | From enrollment to the end of treatment at 1 month
  used to measure the divergent Association ability
Score on the Wsiconsin Card Sorting Test (WCST) | From enrollment to the end of treatment at 1 month
  Used to measure cognitive flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaanxi Provincial Chang'an Compulsory Isolation Drug Rehabilitation Center, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
This study is a government-collaborative project involving sensitive personal information of a vulnerable population, and as such, it is imperative to adhere to strict confidentiality protocols. All data collected will be handled in compliance with ethical guidelines and legal requirements to ensure the protection of participants' privacy.